CLINICAL TRIAL: NCT04127760
Title: A Multicenter Randomized Controlled Trial of the Efficacy of Postoperative Radiotherapy for Atypical Meningioma Without Venous Sinus Invasion After Gross-total Resection
Brief Title: Efficacy of Postoperative Radiotherapy for Atypical Meningioma Without Venous Sinus Invasion After Gross-total Resection
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Collaborators: Sir Run Run Shaw Hospital (Other); Zhejiang Provincial People's Hospital (Other); Ningbo Medical Center Lihuili Hospital (Other Government); Jinhua Central Hospital (Other); Taizhou Hospital (Other); Shaoxing Hospital of Zhejiang University (Other); People's Hospital of Quzhou (Other); Huzhou Central Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ns20191111
Record Dates: First submitted 2019-10-14; First posted 2019-10-16 (Actual); Last update posted 2019-10-16 (Actual); Status verified 2019-10

CONDITIONS: Meningioma Atypical; Radiotherapy; Progression-Free Survival; Adverse Effect of Radiation Therapy
Keywords: Meningioma Atypical; radiotherapy
MeSH Terms: conditions — Radiation Injuries | interventions — Radiotherapy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control (No Intervention): Follow-up at several time frames
- treatment (Experimental): Radiotherapy would be carried out. Follow-up at the same time frames as the control arm
  Interventions: Radiation: radiotherapy

INTERVENTIONS:
Radiation: radiotherapy — Radiotherapy would start within 2 months after the operation, and 5 days of radiotherapy is performed every week. The dose of each radiotherapy is 1.8 Gy for 6 weeks, and the total dose is 54 Gy.
  Arms: treatment

SUMMARY:
Postoperative adjuvant radiotherapy is a key component of comprehensive treatment of meningioma. However, for atypical meningioma after total resection, there is still a huge controversy in patients who need adjuvant radiotherapy after surgery.

Many scholars have focused on this problem and carried out some small-scale retrospective studies, but they have contradictory results. Some of the studies found that postoperative adjuvant radiotherapy could not improve the prognosis of patients, but was questioned because the sample size was too small, resulting in insignificant results, while other studies found that postoperative adjuvant radiotherapy can improve progression free survival. A study based on the National Cancer Database found that postoperative adjuvant radiotherapy and gross tumor resection are associated with a good prognosis. A recent meta-analysis enrolled a total of 757 patients and found that postoperative adjuvant radiotherapy reduced the risk of tumor recurrence but did not improve survival time. Our team reviewed the meningioma data in the SEER database and conducted a study previously. The study found that postoperative adjuvant radiotherapy did not improve the overall survival of these patients. The relevant research results were recently published in Frontiers in oncology. We further reviewed and summarized the single-center data of our hospital and found that postoperative adjuvant radiotherapy could not improve the progression free survival and overall survival of patients. Besides, we also performed a meta-analysis and found that postoperative adjuvant radiotherapy had a trend to improve progression-free survival, but there was no statistical difference.

Because there are many deficiencies in previous researches, and the research results are also contradictory, it is still unclear whether patients with atypical meningioma who have undergone gross total resection can benefit from postoperative adjuvant radiotherapy. Further high quality clinical trials is still needed to be conducted in order to guide the postoperative care of patients. Therefore, we intend to conduct this multicenter randomized controlled trial to determine the value of postoperative adjuvant radiotherapy in patients with atypical meningioma who underwent gross total resection.

DETAILED DESCRIPTION:
The study aims to enroll a total of 140 participants. Subjects would be enrolled with the following information: name, age, gender, contact, KPS score, preoperative ASA score, current ECOG score, tumor location, date of surgery, degree of tumor resection (modified Simpson grade), pathology type, Ki-67 Proliferation index, etc. The preoperative magnetic resonance image of the subject is stored. Tissue specimens are genetically examined.

Using a simple randomization method and random assignment in a 1:1 ratio, a random sequence was first generated, and SAS version 9.1 statistical software was used to generate an allocation sequence table including subject numbers, 140 random numbers, and random groupings. 140 Subjects would be assigned to the test group (n=70) and the control group (n=70) in a 1:1 ratio. The table of the assignment sequence is duplicated and saved by the neurosurgical secretary and the trial designer of the Second Affiliated Hospital of Zhejiang University. The secretary puts the group mark into the 140 opaque kraft envelopes with the serial number 1 to 140 according to the order of the allocation sequence table, and submits them to the test designer. Zhige Guo is responsible for enrolling the participants according to the inclusion criteria, assigning the subjects numbers according to the order of the treatment, and Qiang Zeng is responsible for disassembling the corresponding opaque envelopes according to the number of the subjects, and exerting interventions according to the group marks. Chenhan Ling is responsible for follow-up and regular measurement of various indicators, and Fei Dong is responsible for the images reports. Until the end of the trial, Zhige Guo, Chenhan Ling and Fei Dong would not know the grouping of the subjects.

The test level of the study was α=0.05, and the two-sided test was used. All statistical analysis was performed by SPSS 16.0 statistical software.

1. For PFS, OS, and DSS data, the COX proportional hazards model was used to calculate the hazard ratio (HR) of radiotherapy and to assess the statistical difference between the corresponding prognostic data between the two groups.
2. For the 3-year progression-free survival, 3-year survival rate, and 5-year progression-free survival, 5-year survival rate data, the chi-square test was used to compare the differences between the two groups.

ELIGIBILITY:
Inclusion Criteria:

* Patients who underwent gross total resection at each center and were diagnosed as atypical meningioma (WHO class II) according to the WHO 2016 diagnostic criteria.
* Gross total resection was defined as modified Simpson 1-3 and confirmed by postoperative magnetic resonance imaging.

Exclusion Criteria:

* age less than 18 years old or older than 70 years
* meningioma recurrence
* patients had previous radiotherapy
* multiple meningioma
* optic nerve sheath meningioma or other extracranial meningioma
* tumor involving venous sinus
* ECOG score ≥ 2 points
* preoperative ASA grade ≥ 3
* previous or current malignant tumors
* pregnant or lactating women
* Patients with Gd-DTPA allergies, spatial claustrophobia or pacemaker implantation that can not be conducted constract-enhanced head magnetic resonance examination
* patients who were unable to obtain informed consent or refused to participate in the study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2020-01-01 (Estimated); Primary Completion 2028-01-01 (Estimated); Study Completion 2033-01-01 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival | 60months
  the length of time during and after medication or treatment during which the disease being treated does not get worse

SECONDARY OUTCOMES:
3-year survival rate | 36months
  the percentage of people in a study or treatment group still alive for 3 years after diagnosis
3-year progression-free survival | 36months
  3 years during and after medication or treatment during which the disease being treated does not get worse
5-year survival rate | 60months
  the percentage of people in a study or treatment group still alive for 5 years after diagnosis
10-year progression-free survival | 120 months
  10 years during and after medication or treatment during which the disease being treated does not get worse
10-year survival rate | 120 months
  the percentage of people in a study or treatment group still alive for 10 years after diagnosis
Disease-specific survival | from diagnosis up to 10 years
  the percentage of people in a study or treatment group who have not died from a specific disease in a defined period of time. The time period usually begins at the time of diagnosis or at the start of treatment and ends at the time of death. Patients who died from causes other than the disease being studied are not counted in this measurement
overall survival | from diagnosis up to 10 years
  From randomization to death due to any cause

IPD SHARING:
Plan to Share IPD: No